CLINICAL TRIAL: NCT04471402
Title: Determining the Pharmacogenetic Basis of Non-responsiveness to the Sedative Effects of Dexmedetomidine in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Kong Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Precedex PG study
Record Dates: First submitted 2020-07-08; First posted 2020-07-15 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-08

CONDITIONS: Pharmacogenetic Study; Procedural Anxiety; Dexmedetomidine
Keywords: Procedural anxiety in children; Pharmacogenetic study; Dexmedetomidine; Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swab samples are taken from subjects for DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects recruited: All subjects recruited will be given 3mcg/kg intranasal Precedex through an atomiser, divided equally between two nostrils. They will be observed and sedation score will be recorded every 5 minutes according to the University of Michigan Sedation Scale (UMSS). Pulse oximetry and Blood pressure cuff will be applied whenever they accept these monitoring.
  A buccal swab sample will be taken from all children and the identified genes will be analysed and compared between the different responders (fast, normal, slow or non-responders).
  Interventions: Drug: Precedex

INTERVENTIONS:
Drug: Precedex — Intranasal Precedex 3mcg/kg
  Other Names: Dexmedetomidine

SUMMARY:
Intranasal Dexmedetomidine is one of the sedative drugs of choice commonly used as an anxiolytic premedication for children for diagnostic or therapeutic procedures. However, some children do not achieve the level of sedation expected with the usual dose after an expected timeframe, leading to distress and costly time wasted.

In this study, we would try to identify a genetic basis to non-responders of Dexmedetomidine by comparing a chosen gene panel of 250 relevant genes between responders and non-responders to a standardized 3mcg/kg intranasal Dexmedetomidine.

DETAILED DESCRIPTION:
For most children, having to endure a diagnostic or therapeutic procedure in a hospital environment is a frightening and distressing experience, especially if it is accompanied by pain or discomfort. In an attempt to minimise the trauma and to maximise co-operation from the child, administration of a sedative is often requested by either the parent or the proceduralist. Some sedative agents may have the side effect reducing the child's efforts in breathing, causing inadequate oxygen to be delivered to and carbon dioxide removed from the body, a state that can be life threatening if left untreated. Other sedative agents may cause unpleasant sensations such as hallucinations or nausea while still others may have a paradoxical effect of exciting rather than sedating the child. Among the available agents that may be administered without the presence of an attendant anaesthesiologist, dexmedetomidine is an agent of choice with minimal incidence of the aforementioned effects. However, we have observed in a small proportion of children that dexmedetomidine does not see to be able to elicit a sedative response in the expected time and with the usual dose. It is possible that there is a genetic bas to this resistance and it would be of great use to be able to predict the non-responders ahead of time so an appropriate alternative may be selected without a trial and error approach.

In this project, children who would require Precedex as first-line sedation for radiological or pre-anaesthesia sedation are asked to participate by providing a buccal swab sample and have their genome (genetic makeup) characterised by target sequencing. They are standardized into receiving 3mcg/kg intranasal Precedex and are observed every 5 minutes afterwards for their level of sedation. They would be identified as 'fast responder', 'normal responder', 'slow responder' and 'definite non-responder'.

A gene panel of 250 relevant genes is chosen and compared between the different groups of responders and non-responders. We will then try to look for the differences between these groups and we will use this information to build a predictive model. This model will help to identify non-responders in the future and this would allow clinicians to prepare for an alternative approach to sedation. This would save time, distress to the child and parent and ultimately cost to the institution.

ELIGIBILITY:
Inclusion Criteria:

* Children who would receive 3mcg/kg intranasal Precedex as a first line sedative agent for radiological procedures or for pre-anaesthesia sedation
* Written informed consent from parent or legal guardian

Exclusion Criteria:

* Known allergy or hypersensitivity to Precedex
* Pre-existing developmental delay
* Neurological impairment
* Autism
* Fever (temperature >/= 38.5c)
* Major organ dysfunction
* Cardiac arrhythmia
* Cardiac failure
* Subjects who would require a dose exceeding 100mcg if 3mcg/kg dose is achieved
* Subjects who have failed intranasal administration of Dexmedetomidine

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who require intranasal Precedex at 3 mcg/kg as an anxiolytic premedication for radiological or pre-anaesthesia sedation in Hong Kong Children's Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sedative response to intranasal Precedex | Every 5 minutes till 30 minutes from administration of intranasal Precedex
  Sedation response is recorded every 5 minutes after administration of Precedex until a satisfactory sedation level is reached. A satisfactory sedation level is defined as a UMSS of 3-4 (University of Michigan Sedation Scale) and allowing transfer to bed without waking up. Subjects are categorized into 'fast responder', 'normal responder', 'slow responder' and 'definite non-responder' based on the time required to achieve satisfactory level of sedation

SECONDARY OUTCOMES:
Onset time of sedation | 45 minutes from administration of intranasal Precedex
  The actual time required to reach a satisfactory sedation level after administration of intranasal Precedex
Incidence of bradycardia | 2 hour from administration of intranasal Precedex or until administration of other sedative or anaesthetic drugs, whichever is shorter
  Defined as more than 20% reduction in heart rate from baseline or from the lower limit of published normal values for age, whichever is lower
Incidence of hypotension | 2 hours from administration of intranasal Precedex, or until administration of other sedative or anaesthetic drugs, whichever is shorter
  Defined as a systolic blood pressure more than 20% lower than the published normal values for age
Incidence of hypertension | 2 hours from administration of intranasal Precedex, or until administration of other sedative or anaesthetic drugs, whichever is shorter
  Defined as a systolic blood pressure more than 20% higher than the published normal values for age
Incidence of hypoxia | 2 hours from administration of intranasal Precedex, or until administration of other sedative or anaesthetic drugs, whichever is shorter
  Defined as a SpO2 < or equal to 93% or more than 5% decrease from baseline
Wake up time | 1 hour after completion of procedure
  Time to reach UMSS of 1 or below after completion of procedure
Length of procedure | 3 hours
  Length of procedure is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Vivian MY Yuen, M.D., Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No